CLINICAL TRIAL: NCT03754491
Title: Division of Hepato-gastroenterology; Department of Internal Medicine, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung,Taiwan
Brief Title: The Comparisons of One-stage Stone Removal in Mild and Moderate Cholangitis
Acronym: ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gimy54861439
Record Dates: First submitted 2018-10-15; First posted 2018-11-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-02

CONDITIONS: Cholangitis; Choledocholithiasis
Keywords: Acute cholangitis; choledocholithiasis; ERCP; One-stage treatment
MeSH Terms: conditions — Cholangitis; Choledocholithiasis

STUDY DESIGN:
Intervention Model Description: Investigators will enroll 204 naïve papilla with a body temperature ≥37 °C who was diagnosed with mild or moderate cholangitis associated with choledocholithiasis for one-stage procedure to remove CBD stone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One stage stone removal in mild cholangitis (Experimental): one-stage stone removal at the first session of ERCP in mild cholangitis patients. The indomethacin 100mg anal route will be administered for all patients without allergy history
  Interventions: Behavioral: One stage treatment for mild and moderate cholangitis with choledocholithiasis
- One stage stone removal in moderate cholangitis (Experimental): one-stage stone removal at the first session of ERCP in moderate cholangitis patients. The indomethacin 100mg anal route will be administered for all patients without allergy history
  Interventions: Behavioral: One stage treatment for mild and moderate cholangitis with choledocholithiasis

INTERVENTIONS:
Behavioral: One stage treatment for mild and moderate cholangitis with choledocholithiasis — one stage of stone removal in mild or moderate cholangitis.

SUMMARY:
In expert comment, performing the sphincterotomy for choledocholithiasis with acute cholangitis may increase bleeding and pancreatitis risks (from 2% to 10%). Therefore, investigators often perform biliary drainage in acute stage, and arrange 2nd session ERCP for stone removal later. However, in the recent study, single-stage endoscopic treatment may be still effective (stone removal rate 90%) and safe for mild to moderate acute cholangitis associated with choledocholithiasis. Investigators will carry out a prospective trial to analyze one-stage retrograde endoscopic common bile duct stone removal in mild and moderate cholangitis with choledocholithiasis to determine the safety, successful rate, and complications in these two groups.

DETAILED DESCRIPTION:
Investigators will enroll 204 naïve papilla with a body temperature ≥37 °C who was diagnosed with mild to moderate cholangitis associated with choledocholithiasis. The method of one-stage: performing the stone removal at the first session of ERCP. The pancreas duct stent will be placed for preventing post ERCP pancreatitis (PEP) if necessary. The indomethacin 100mg anal route will be administered for all patients without allergy history. All participants will receive the empiric antibiotics treatment for cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* naïve papilla with a body temperature ≥37 °C who was diagnosed with mild to moderate cholangitis associated with choledocholithiasis.

Exclusion Criteria:

* procedural failure requiring an anatomy-modifying procedure, such as a Billroth II subtotal gastrectomy or R-en-Y gastrojejunostomy ;
* stenosis of the pyloric ring ;
* tumor-related obstruction;
* failure to locate the papilla ;
* active peptic ulcer bleeding ;
* intolerance due to inadequate sedation
* CBD sludge;
* non-naïve papilla in ERCP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Post ERCP pancreatitis | After ERCP, an average of 7 days
  Serum amylase > 3 times of (115 IU/L) with clinical abdominal pain
Bowel perforation | After ERCP, an average of 7 days
  Participants with sign of bowel perforation after ERCP
Papillary bleeding | After ERCP, an average of 7 days
  Participants with papillary bleeding after ERCP
Success rate of stone removal | an average of 14 days.
  Complete bile duct stone clearance
Cost of hospitalization | From emergent department to the timing of being discharged, and an average of 30 days
  Total cost in two individual groups in hospitalization.

SECONDARY OUTCOMES:
Mortality | an average of 30 days
  Mortality during and after discharged

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-MING LIANG, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miura F, Takada T, Strasberg SM, Solomkin JS, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Yoshida M, Mayumi T, Okamoto K, Gomi H, Kusachi S, Kiriyama S, Yokoe M, Kimura Y, Higuchi R, Yamashita Y, Windsor JA, Tsuyuguchi T, Gabata T, Itoi T, Hata J, Liau KH; Tokyo Guidelines Revision Comittee. TG13 flowchart for the management of acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):47-54. doi: 10.1007/s00534-012-0563-1. PMID 23307003
- [Result] Eto K, Kawakami H, Haba S, Yamato H, Okuda T, Yane K, Hayashi T, Ehira N, Onodera M, Matsumoto R, Matsubara Y, Takagi T, Sakamoto N; Hokkaido Interventional EUS/ERCP study (HONEST) group. Single-stage endoscopic treatment for mild to moderate acute cholangitis associated with choledocholithiasis: a multicenter, non-randomized, open-label and exploratory clinical trial. J Hepatobiliary Pancreat Sci. 2015 Dec;22(12):825-30. doi: 10.1002/jhbp.296. Epub 2015 Nov 25. PMID 26510180
- [Derived] Liang CM, Chiu YC, Lu LS, Wu CK, Sou FM, Chiu SM, Lee YC, Huang PY, Chuah SK, Kuo CM. Early and Direct Endoscopic Stone Removal in the Moderate Grade of Acute Cholangitis with Choledocholithiasis Was Safe and Effective: A Prospective Study. Life (Basel). 2022 Nov 30;12(12):2000. doi: 10.3390/life12122000. PMID 36556365